CLINICAL TRIAL: NCT04481906
Title: Long-term Follow-up of Vaginal Mesh Procedures for Female Cystocele
Brief Title: Vaginal Mesh Procedures for Female Cystocele
Status: Completed | Type: Observational
Sponsor: Cathay General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CGH-P100072
Record Dates: First submitted 2018-07-16; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2018-07

CONDITIONS: Cystocele
Keywords: cystocele; pelvic floor muscle exercise; anterior vaginal repair; vaginal mesh
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Women 20 years and older with cystocele: Women 20 years and older with cystocele
  Interventions: Procedure: Vaginal mesh for female cystocele

INTERVENTIONS:
Procedure: Vaginal mesh for female cystocele — Vaginal mesh procedures (e.g. Perigee) were susgested for women with POP-Q stage III or more cystocele

SUMMARY:
This study aimed to evaluate primarily the functional outcomes and secondly the morphological outcomes for women who had received standard managements for cystocele at mediate-term follow-up.

DETAILED DESCRIPTION:
Pelvic organ prolapsed (POP) is an important health issue for women all over the world, with cystocele being the commonest type of POP. The side effects related to cystocele include voiding dysfunction, urinary retention, urinary tract infection, hydroureter, or hydronephrosis. The management for cystocele can be classified as non-surgical and surgical methods. Non-surgical methods comprise pelvic floor muscle exercise and vaginal pessaries, while surgical methods can be divided as conventional operations and operations applying mesh augmentation. Conventional surgeries for cystocele such as anterior colporrhapy have high surgical failure rates and complications including vaginal shortening or vaginal stenosis. Operations applying mesh augmentation are becoming the mainstream in the surgeries for cystocle. The Perigee System (American Medical Systems, Minnetonka, MN, USA), which has been approved by American FDA and Taiwan DOH in treating female cystocele, have promising short-term surgical outcomes. However, long-term reports incorporating both functional and morphological outcomes are lacking in the literatures. This study aimed to evaluate primarily the functional outcomes and secondly the morphological outcomes for women who had received standard managements for cystocele at mediate-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cystocele

Exclusion Criteria:

* Pregnancy or possibility of future pregnancy
* Urinary tract infection
* Diabetes
* Neurological diseases
* Cardiovascular diseases

Min Age: 240 Months | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women 20 years or older with cystocele
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2011-10-25; Primary Completion 2012-06-16 (Actual); Study Completion 2014-10-05 (Actual)

PRIMARY OUTCOMES:
POP-Q Ba point | Preoperative, as well as postoperative 3 months, 12 months, and then anuuanlly
  POP-Q Ba > II POP-Q stage

SECONDARY OUTCOMES:
Functional and ultrasound manifestations | Preoperative, as well as postoperative 3 months, 12 months, and then anuuanlly
  Urinary incontinence, overactive bladder symptoms, voiding dysfunction, bladder neck position on ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Cathay General Hospital, Taipei, Taiwan